CLINICAL TRIAL: NCT00945919
Title: A Pilot Study of Ultra Rapid Opioid Rotation and Titration of Oxymorphone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Marco Pappagallo, MD, Director of Pain Research and Development, Mount Sinai School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO# 08-1423
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Nociceptive Pain; Neuropathic Pain; Non-cancer Pain
Keywords: Oral morphine; oxycodone; OPANA; Oxymorphone; pain; nociceptive; neuropathic; rotation; titration; mixed origin non-cancer pain
MeSH Terms: conditions — Neuralgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxymorphone ER — Rapid Opioid rotation/titration

SUMMARY:
This project will explore the safety and feasibility of performing a successful intravenous patient controlled analgesia (IV PCA) Oxymorphone titration and conversion to oral ER Oxymorphone (extended release or OPANA ER) in the outpatient setting.

DETAILED DESCRIPTION:
This project will enroll 12 volunteers who suffer from chronic pain. Potential participants must be on one of the following therapies:

* Long acting morphine
* Oxycodone Participants will be asked to complete a pain diary for approximately 10 days and to stop taking their current pain medications the night before they are admitted o the GCRC. Once the patients present at the GCRC, they will be started on the IV PCA (Patient Controlled Analgesia) Oxymorphone to control their pain. Titration will take approximately a total of 8 hrs. At the end of the titration period, patients will be discharged home on OPANA ER. The oral dose will be calculated based on the IV PCA use. During the titration, patients' pain, vital and side effects will be assessed hourly until the 8th hour of the IV PCA titration.

Patients will be contacted daily by a member of the study team to assess pain and side effects. The OPANA ER dose will be adjusted as needed to adequately manage both.

If patients do not feel as though they are getting adequate pain relief, they can return to their previous medication, at which point they are considered withdrawn from the study.

Patients will undergo an exit examination 2 weeks after they were admitted to the GCRC in order to assess pain relief. In addition, a final follow-up telephone interview will take place 6 weeks after the initial 1-day stay at the GCRC. Our research staff or physicians will ask about your pain treatment and ask which Opioid medication you are currently taking.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Chronic pain of nociceptive, neuropathic, or mixed origin.
* Patients with chronic non-cancer pain.
* Ongoing chronic Opioid treatment with either oral morphine or oxycodone (long term-more than three months and at least a total daily Opioid dose of 60mg morphine or of 30 mg oxycodone).
* Pain of moderate intensity (>= 4, on the numerical scale 0-10) despite ongoing Opioid therapy.
* Non-pregnant, non-lactating women.
* Sufficient language skills to communicate with research staff.

Exclusion Criteria:

* Non-ambulatory patients.
* Clinically significant respiratory, renal, hepatic, or cardiac disease.
* Documented diagnosis of sleep apnea (the study physician may exclude patients who present with clinical features and complaints suggestive of a diagnosis of probably sleep apnea).
* History of illicit drug or alcohol dependence or abuse, abnormal drug taking/seeking behaviors.
* Sever depression (> 26 on the BDI) or severe anxiety or insomnia requiring chronic daily use of benzodiazepines or hypnotic drugs.
* Patients who exhibit a score on the Mini Mental Status Exam (MMSE) of 26 or less. (The range of scores for mild dementia is 21-26 on the MMSE).
* Hypersensitivity to study medication (Oxymorphone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The safety of rapid Opioid rotation | Daily for two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States